CLINICAL TRIAL: NCT00890019
Title: A Phase I Study to Assess the Safety and Immunogenicity of New Malaria Vaccine Candidate AdCh63 ME-TRAP, Alone and With MVA ME-TRAP, Using a Prime-boost Delivery Schedule
Brief Title: A Study of AdCh63 ME-TRAP Alone and With MVA ME-TRAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC033
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1A, 2A, 3A, 4A, 5A, 6A, 7A (Experimental): AdCh63 ME-TRAP
  Interventions: Biological: AdCh63 ME-TRAP
- 1B, 2B, 3B, 4B, 6B, 7B, 7C (Experimental): AdCh63 ME-TRAP; MVA ME-TRAP
  Interventions: Biological: AdCh63 ME-TRAP; MVA ME-TRAP

INTERVENTIONS:
Biological: AdCh63 ME-TRAP — 1. A:Intradermal injection 1x10^8 vp at day 0
  2. A:Intradermal injection 1x10^9 vp at day 0
  3. A:Intradermal injection 1x10^10 vp at day 0
  4. A:Intradermal injection 5x10^10 vp at day 0
  5:Intramuscular injection 1x10^10 vp at day 0
  6A:Intramuscular injection 5x10^10 vp at day 0
  7A: Intramuscular injection 2x10^11 vp at day 0
  Other Names: Simian adenovirus expressing P. falciparum antigens ME-TRAP
  Arms: 1A, 2A, 3A, 4A, 5A, 6A, 7A
Biological: AdCh63 ME-TRAP; MVA ME-TRAP — 1. B: AdCh63 ME-TRAP intradermally at dose of 1x10^8 vp at day 0; MVA ME-TRAP intradermally at dose of 2x10^8 pfu at day 56 (+/- 7 days)
  2. B: AdCh63 ME-TRAP intradermally at dose of 1x10^9 vp at day 0; MVA ME-TRAP intradermally at dose of 2x10^8 pfu at day 56 (+/- 7 days)
  3. B: AdCh63 ME-TRAP intradermally at dose of 1x10^10 vp at day 0; MVA ME-TRAP intradermally at dose of 2x10^8 pfu at day 56 (+/- 7 days)
  4. B: AdCh63 ME-TRAP intradermally at dose of 5x10^10 vp at day 0; MVA ME-TRAP intradermally at dose of 2x10^8 pfu at day 56 (+/- 7 days)
  6B: AdCh63 ME-TRAP intramuscularly at dose of 5x10^10 vp at day 0; MVA ME-TRAP intradermally at dose of 2x10^8 pfu at day 56 (+/- 7 days)
  7B and 7C: AdCh63 ME-TRAP intramuscularly at dose of 2x10^11 vp at day 0; MVA ME-TRAP intradermally at dose of 2x10^8 pfu at day 56 (+/- 7 days)
  Other Names: Simian adenovirus, modified vaccinia Ankara virus
  Arms: 1B, 2B, 3B, 4B, 6B, 7B, 7C

SUMMARY:
This is an open label phase I study, to assess the safety of a novel malaria vaccine, AdCh63 ME-TRAP, simian adenovirus encoding Plasmodium falciparum antigens. This follows promising phase I clinical studies of MVA ME-TRAP and preclinical studies of AdCh63 and MVA ME-TRAP used together in prime-boost regimes. All volunteers recruited will be healthy adults. They will be primed with various doses of AdCh63 ME-TRAP administered intradermally or intramuscularly. Some of the volunteers will receive a booster vaccination with MVA ME-TRAP at various doses administered via the intradermal or intramuscular route. Safety data will be collected for each of the eight regimens. Secondary aims of this study will be to assess the immune responses generated by each of these regimes.

DETAILED DESCRIPTION:
ME-TRAP insert contains a fusion protein of multiple epitopes (ME) and the Plasmodium falciparum pre-erythrocytic thrombospondin-related adhesion protein (TRAP). The 'ME' is a string of 20 epitopes fused to the thrombospondin-related adhesion protein. TRAP was selected as it is well characterized and has a protective homologue in rodents. We have safely administered ME-TRAP to over 700 volunteers in the UK and Africa.

MVA vector proved to be non-contagious and avirulent. Viral replication is blocked late during infection of cells but importantly viral and recombinant protein synthesis is unimpaired even during this abortive infection. Replication-deficient recombinant MVA has been viewed as an exceptionally safe viral vector. When tested in animal model studies recombinant MVAs have been shown to be avirulent, yet protectively immunogenic as vaccines against viral diseases and cancer. Recent studies in macaques severely immuno-suppressed by SIV infection have further supported the view that MVA should be safe in immuno-compromised humans.

Simian adenoviruses have not been used previously in a clinical trial in humans. However, they are under active development as vaccines for HIV, (by GSK), and for HCV, (Merck).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* Willing to use barrier contraception until three months after the last vaccination
* For females only negative pregnancy test on the day(s) of vaccination
* Agreement to refrain from blood donation during the course of the study
* Written informed consent

Exclusion Criteria:

* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of a recombinant MVA vaccine containing a relevant antigen (for those in B groups) or adenoviral vaccine, (all volunteers).
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products, Kathon.
* History of clinically significant contact dermatitis
* Any history of anaphylaxis in reaction to vaccination
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Seropositive for simian adenovirus 63 (antibodies to AdCh63) at a titre >1 ;200
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* Any other significant disease, disorder or finding, which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or may influence the result of the study, or the volunteer's ability to participate in the study.
* Any history of malaria or
* Travel to a malaria endemic region during the study period or within the previous six months
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
* Any other finding which in the opinion of the investigators would significantly increase the risk of having an adverse outcome from participating in the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2007-07; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To assess the safety of a new malaria vaccine, AdCh63 ME-TRAP, when administered individually and sequentially with MVA ME-TRAP in a prime-boost regime to healthy volunteers | 24 months

SECONDARY OUTCOMES:
To assess the cellular immune response generated, and whether this is affected by immunity to human adenovirus, by AdCh63 ME-TRAP when administered individually and sequentially with MVA ME-TRAP in a prime-boost regime to healthy volunteers | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, Professor, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Lister Ward, Department of Infection and Tropical Medicine, Northwick Park Hospital, Harrow, Middlesex
  - Oxford Vaccine Group, Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Churchill Hospital, Oxford, Oxfordshire

REFERENCES:
- [Derived] O'Hara GA, Duncan CJ, Ewer KJ, Collins KA, Elias SC, Halstead FD, Goodman AL, Edwards NJ, Reyes-Sandoval A, Bird P, Rowland R, Sheehy SH, Poulton ID, Hutchings C, Todryk S, Andrews L, Folgori A, Berrie E, Moyle S, Nicosia A, Colloca S, Cortese R, Siani L, Lawrie AM, Gilbert SC, Hill AV. Clinical assessment of a recombinant simian adenovirus ChAd63: a potent new vaccine vector. J Infect Dis. 2012 Mar 1;205(5):772-81. doi: 10.1093/infdis/jir850. Epub 2012 Jan 24. PMID 22275401